CLINICAL TRIAL: NCT02630823
Title: Immunotherapy With MK-3475 in Surgically Resectable Endometrial Carcinoma
Brief Title: MK-3475 Immunotherapy in Endometrial Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201601062
Record Dates: First submitted 2015-12-10; First posted 2015-12-15 (Estimated); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Endometrial Cancer; Endometrial Carcinoma; Neoplasms, Endometrial
MeSH Terms: conditions — Endometrial Neoplasms | interventions — pembrolizumab; Standard of Care; Paclitaxel; Carboplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1: MK-3475 (Experimental): * Patients will undergo endometrial biopsy followed by 2 doses of MK-3475 3 weeks apart. 3-4 weeks after the second dose of MK-3475, the standard of care surgical resection will take place, followed by standard of care adjuvant therapy. Tissue and blood will be collected at the time of surgical resection for immune analysis. For patients whose pathology confirms high-risk features and advanced stage, MK-3475 will be given every 3 weeks starting 4 -6 weeks after completion of adjuvant therapy for a maximum of 4 doses post-surgery.
  * MK-3475 will be given intravenously at a dose of 200 mg over the course of 30 minutes.
  * The standard of care chemotherapy will consist of 6 cycles of paclitaxel and carboplatin AUC 5 every 3 weeks for 6 cycles.
  * The decision to administer radiation therapy will be per the treating physician. If the patient does not receive radiation therapy, then the patient will start MK-3475 every 3 weeks x 4 doses after the completion of chemotherapy.
  Interventions: Drug: MK-3475; Procedure: Surgical resection (standard of care); Drug: Paclitaxel (standard of care); Drug: Carboplatin (standard of care); Radiation: Radiation (standard of care); Procedure: Endometrial biopsy; Procedure: Peripheral blood draw

INTERVENTIONS:
Drug: MK-3475
  Other Names: pembrolizumab; Keytruda
Procedure: Surgical resection (standard of care)
Drug: Paclitaxel (standard of care)
  Other Names: Taxol
Drug: Carboplatin (standard of care)
  Other Names: Paraplat; Paraplatin
Radiation: Radiation (standard of care)
Procedure: Endometrial biopsy
Procedure: Peripheral blood draw

SUMMARY:
Due to the high expression of PD-L1 in endometrial cancers as well as in ovarian cancers which are molecularly similar to uterine serous cancers, using pembrolizumab should be beneficial in this patient population. Since the investigators are able to get a pre-treatment research- related endometrial biopsy as well as the surgical specimen post two cycles of pembrolizumab, the investigators will be able to evaluate the mechanism of action of this drug on the endometrial cancer tumor environment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FIGO grade 3 endometrioid cancer, serous, clear cell, or mixed high grade endometrial cancer with confirmation on research-related endometrial biopsy.
* Radiographically confirmed endometrial adenocarcinoma of stages III-IV requiring adjuvant therapy. If stage III disease is suspected, there should be multiple pelvic and/or lymph nodes involved.
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >10 mm with CT scan, as >20 mm by chest x-ray, or >10 mm with calipers by clinical exam by RECIST 1.1.
* Treatment plan must include primary site biopsy followed by resection of the primary tumor site and any metastatic sites at time of surgery.
* At least 18 years of age.
* GOG performance status ≤ 2
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl
  * Hemoglobin ≥ 9 g/dL
  * Total bilirubin ≤ 1.5 x IULN OR direct bilirubin ≤ IULN for patients with total bilirubin > 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN (or ≤ 5 x IULN for patients with liver metastases)
  * Serum creatinine ≤ 1.5 x IULN OR creatinine clearance by Cockcroft-Gault ≥ 60 mL/min/1.73 m2 for patients with creatinine levels > 1.5 x IULN
  * INR or PT ≤ 1.5 x IULN unless patient is receiving anticoagulant therapy as long as INR or PTT is within therapeutic range of intended use of anticoagulants
  * aPTT ≤ 1.5 x IULN unless patient is receiving anticoagulant therapy as long as INR or PTT is within therapeutic range of intended use of anticoagulants
* Sexually active women of childbearing potential must agree to contraceptive methods as described by the protocol prior to study entry, for the duration of pre-operative study participation and until definitive hysterectomy/bilateral salpingo-oophorectomy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* FIGO grade 1 or 2 endometrioid cancer.
* Radiographic imaging demonstrating uterine cancer that is probably stage I or II.
* Prior treatment for endometrial cancer.
* Prior treatment with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to first dose of MK-3475 or has not recovered (i.e., to ≤ grade 1 or baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to the first dose of MK-3475 or has not recovered (i.e., to ≤ grade 1 or baseline) from adverse events due to a previously administered agent. Note, subjects with ≤ grade 2 neuropathy are an exception to this criterion and may qualify for the study. Note, if a subject received major surgery, she must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Received a live vaccine within 30 days prior to the first dose of MK-3475. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. FluMist) are live attenuated vaccines and are not allowed.
* A history of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only.
* Known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of MK-3475 and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy in dosing exceeding 10 mg daily of prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of MK-3475.
* Currently receiving any other investigational agents or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of MK-3475.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-3475 or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring systemic therapy, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, immunosuppression, autoimmune conditions, underlying pulmonary disease, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Pregnant and/or breastfeeding. Patient must have a negative serum or urine pregnancy test within 72 hours of study entry.
* Known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as HCV RNA [qualitative] is detected).
* Known history of HIV (HIV 1/2 antibodies).
* Known history of active TB.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02-05 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Premal Thaker, M.D., MSc., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: MK-3475
Started | 10
Completed | 8
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Did not undergo cytoreductive surgery due to pre-operative disease progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1: MK-3475
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 60 [46 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Safety as Measured by Any Grade Treatment Related Adverse Events Experienced by ≥ 2 Patients
Description: -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all adverse event reporting
Time Frame: Through 90 days following last dose of MK-3475 (approximately 56 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: MK-3475
Number analyzed (Participants) | 10
Participants
  Abdominal pain | 10
  Nausea | 9
  Constipation | 8
  Cough | 8
  Dyspnea | 8
  Peripheral neuropathy | 8
  Alopecia | 7
  Fatigue | 7
  Anemia | 6
  Blurred vision | 6
  Depression | 6
  Bloating | 5
  Bruising | 5
  Headache | 5
  Hyperglycemia | 5
  Vaginal hemorrhage | 5
  Vomiting | 5
  Leukocytosis | 5
  Increased ALT | 4
  Anorexia | 4
  Back pain | 4
  Hot flashes | 4
  Hypoalbuminemia | 4
  Myalgia | 4
  Pain in extremity | 4
  Rash acneiform | 4
  Increased alkaline phosphatase | 3
  Chest pain | 3
  Dizziness | 3
  Hypocalcemia | 3
  Hyponatremia | 3
  Neutropenia | 3
  Palpitations | 3
  Rash maculo-papular | 3
  Urinary incontinence | 3
  Limb edema | 3
  Infusion related reaction | 3
  Abdominal distension | 2
  Anxiety | 2
  Increased AST | 2
  Chills | 2
  Dysmenorrhea | 2
  Hearing impaired | 2
  Hematuria | 2
  Hyperkalemia | 2
  Hypokalemia | 2
  Hypothyroid | 2
  Malaise | 2
  Menorrhagia | 2
  Mucositis | 2
  Pain | 2
  Decreased platelets | 2
  Pruritus | 2
  Respiratory, thoracic and mediastinal disorders | 2
  Urinary urgency | 2

2. Primary Outcome: Safety as Measured by Any Grade 3 or Higher Treatment Related Adverse Events
Description: as for outcome 1
Time Frame: Through 90 days following last dose of MK-3475 (approximately 56 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: MK-3475
Number analyzed (Participants) | 10
Participants
  Anemia | 4
  Neutropenia | 3
  Hyperglycemia | 2
  Decreased white blood cells | 2
  Menorrhagia | 1
  Heart failure | 1
  Hypophosphatemia | 1
  Pulmonary edema | 1
  Bone infection | 1

3. Secondary Outcome: Progression-free Survival (PFS)
Description: * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: Up to 2 years following completion of therapy (median follow-up of 35 months (full range 11.3-46 months)
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Arm 1: MK-3475
Number analyzed (Participants) | 10
weeks | 201.3 (160.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment through 30 days following the last day of study treatment and adverse events of clinical interest were followed through 90 days following the last day of study treatment (approximately 56 weeks). All-cause mortality was collected from start of treatment through completion of follow-up (median follow-up of 35 months, full range 11.3-46 months).
Arm/Group | Arm 1: MK-3475
All-Cause Mortality (participants affected / at risk) | 5/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: MK-3475 (N=10)
Congestive heart failure (Cardiac disorders) | 1
Pulmonary pretension (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: MK-3475 (N=10)
Anemia (Blood and lymphatic system disorders) | 6
Chest pain - cardiac (Cardiac disorders) | 3
Palpitations (Cardiac disorders) | 3
Sinus tachycardia (Cardiac disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 2
Vertigo (Ear and labyrinth disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Changes in vision - near sighted (Eye disorders) | 1
Blurred vision (Eye disorders) | 6
Dysgeusia (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 9
Ascites (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 9
Rectal hemorrhage (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Night sweats (General disorders) | 1
Chills (General disorders) | 2
Edema face (General disorders) | 1
Edema limbs (General disorders) | 3
Edema trunk (General disorders) | 1
Fatigue (General disorders) | 7
Fever (General disorders) | 1
Infusion related reaction (General disorders) | 1
Malaise (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 3
Upper respiratory tract infection (Infections and infestations) | 2
Bone infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 5
Wound complication (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 4
Alkaline phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 2
White blood cell decreased (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Paresthesia (Musculoskeletal and connective tissue disorders) | 2
Ankle pain (Musculoskeletal and connective tissue disorders) | 1
Lumps in arms (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Carpal tunnel syndrome (Musculoskeletal and connective tissue disorders) | 2
Cognitive disturbance (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 8
Presyncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 6
Personality change (Nervous system disorders) | 1
Hematuria (Renal and urinary disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 3
Urinary tract pain (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 2
Dysmenorrhea (Reproductive system and breast disorders) | 2
Dyspareunia (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 2
Pelvic pain (Reproductive system and breast disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 5
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 7
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Nail loss (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hot flashes (Vascular disorders) | 4
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/23/NCT02630823/Prot_SAP_000.pdf